CLINICAL TRIAL: NCT04475341
Title: 'A Randomized Clinical Trial on the Clinical Efficacy of Bone Marrow Stimulation Combined With the Insertion of Bone Marrow Aspirate Concentrate (BMAC) for the Treatment of Small Primary and Non-primary Talar Osteochondral Lesions'
Brief Title: Osteochondral Lesions Under 15mm2 of the Talus; is Iliac Crest Bone Marrow Aspirate Concentrate the Key to Success?
Acronym: OUTBACK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jari Dahmen, MD, BSc, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GK2019OUTBACK
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Osteochondral Lesion of Talus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMS without BMAC (Active Comparator)
  Interventions: Procedure: BMS alone
- BMS with BMAC (Experimental)
  Interventions: Biological: BMS + Bone Marrow Aspirate Concentrate

INTERVENTIONS:
Biological: BMS + Bone Marrow Aspirate Concentrate — Both groups of patients are surgically treated with arthroscopic bone marrow stimulation (BMS). The control group will receive BMS alone but with a sham-treatment consisting of a Jamashidi (bone marrow aspiration) needle puncture of the iliac crest. The aspirated bone marrow concentrate will be collected and sent for cell characterisation but will not be inserted in the talar OCD. The intervention group will also receive arthroscopic BMS. From this group, BMAC from the iliac crest will be taken by the same needle puncture. Part of this concentrate will be sent for cell characterisation. Another part will be implanted into the talar OCD.
  Arms: BMS with BMAC
Procedure: BMS alone — Both groups of patients are surgically treated with arthroscopic bone marrow stimulation (BMS). The control group will receive BMS alone but with a sham-treatment consisting of a Jamashidi (bone marrow aspiration) needle puncture of the iliac crest. The aspirated bone marrow concentrate will be collected and sent for cell characterisation but will not be inserted in the talar OCD. The intervention group will also receive arthroscopic BMS. From this group, BMAC from the iliac crest will be taken by the same needle puncture. Part of this concentrate will be sent for cell characterisation. Another part will be implanted into the talar OCD.
  Arms: BMS without BMAC

SUMMARY:
Osteochondral defects (OCDs) of the talus have a significant impact on the quality of life of patients. When OCDs are of small nature (up to 15 mm in diameter), and have failed conservative management, surgical intervention may be necessary. For small cystic defects the current treatment is an arthroscopic bone marrow stimulation (BMS) procedure, during which the damaged cartilage is resected and the subchondral bone is microfractured (MF), in order to disrupt intraosseous blood vessels and thereby introduce blood and bone marrow cells into the debrided lesion, forming a microfracture fibrin clot, which contains a dilute stem cell population from the underlying bone marrow. This procedure has been reported to have a 75% successful long-term outcome. Recently, the additional use of biological adjuncts has become popular, one of them being bone marrow aspirate concentrate (BMAC) from the iliac crest. BMAC consists of mesenchymal stem cells, hematopoietic stem cells and growth factors, which may therefore theoretically improve the quality of subchondral plate and cartilage repair. The current evidence for treating talar OCDs with BMS plus BMAC is limited and heterogeneous. It is unclear to what extent the treatment of talar OCDs with BMS plus BMAC is beneficial in comparison to BMS alone.

DETAILED DESCRIPTION:
Osteochondral defects (OCDs) of the talus have a significant impact on the quality of life of patients. When OCDs are of small nature (up to 15 mm in diameter), and have failed conservative management, surgical intervention may be necessary. For small cystic defects the current treatment is an arthroscopic bone marrow stimulation (BMS) procedure, during which the damaged cartilage is resected and the subchondral bone is microfractured (MF), in order to disrupt intraosseous blood vessels and thereby introduce blood and bone marrow cells into the debrided lesion, forming a microfracture fibrin clot, which contains a dilute stem cell population from the underlying bone marrow. This procedure has been reported to have a 75% successful long-term outcome. Recently, the additional use of biological adjuncts has become popular, one of them being bone marrow aspirate concentrate (BMAC) from the iliac crest. BMAC consists of mesenchymal stem cells, hematopoietic stem cells and growth factors, which may therefore theoretically improve the quality of subchondral plate and cartilage repair. The current evidence for treating talar OCDs with BMS plus BMAC is limited and heterogeneous. It is unclear to what extent the treatment of talar OCDs with BMS plus BMAC is beneficial in comparison to BMS alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a symptomatic OCL of the talus who are scheduled for arthroscopic debridement and microfracture
* OCL depth and/or diameter ≤ 15 mm on computed tomography medial-lateral and/or anterior-posterior
* Age 18 years or older
* Intact remaining articular cartilage of the joint Kellgren-Lawrence stage 0-1

Exclusion Criteria:

* Concomitant OCL of the tibia
* Ankle osteoarthritis grade 2 or 3 van Dijk et al. [53]
* Ankle fracture < 6 months before scheduled arthroscopy
* Inflammatory arthropathy (e.g Rheumatoid arthritis)
* History of (or current) hemopoeitic disease or immunotherapy
* Acute or chronic instability of the ankle
* Use of prescribed orthopaedic shoewear
* Other concomitant painful or disabling disease of the lower limb
* Pregnancy
* Implanted pacemaker
* Participation in previous trials < 1 year, in which the subject has been exposed to radiation (radiographs or CT)
* Patients who are unable to fill out questionnaires and cannot have them filled out
* No informed consent
* HIV positive or hepatitis B or C infection (based on the anamnesis of the patient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-02 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale of Pain During Weightbearing | 2 years post-operatively

SECONDARY OUTCOMES:
EQ5D | pre-operatively
EQ5D | three months postoperatively
EQ5D | one-year post-operatively
EQ5D | two years post-operatively
AOFAS | preoperatively
  American Orthopaedic Foot and Ankle Score (AOFAS)
AOFAS | three months postoperatively
  American Orthopaedic Foot and Ankle Score (AOFAS)
AOFAS | one-year post-operatively
  American Orthopaedic Foot and Ankle Score (AOFAS)
AOFAS | two years post-operatively
  American Orthopaedic Foot and Ankle Score (AOFAS)
FAOS | pre-operatively
  Foot and Ankle Outcome Score
FAOS | three months
  Foot and Ankle Outcome Score
FAOS | one-year post-operatively
  Foot and Ankle Outcome Score
FAOS | two years post-operatively
  Foot and Ankle Outcome Score
NRS in rest | pre-operatively
  Numeric Rating Scale of Pain During Rest
NRS in rest | 3 months postoperatively
  Numeric Rating Scale of Pain During Rest
NRS in rest | 1 year postoperatively
  Numeric Rating Scale of Pain During Rest
NRS in rest | 2 years postoperatively
  Numeric Rating Scale of Pain During Rest
NRS during running | pre-operatively
  Numeric Rating Scale of Pain During Running
NRS during running | 3 months postoperatively
  Numeric Rating Scale of Pain During Running
NRS during running | 1 year postoperatively
  Numeric Rating Scale of Pain During Running
NRS during running | 2 years postoperatively
  Numeric Rating Scale of Pain During Running
NRS during stair-climbing | pre-operatively
  Numeric Rating Scale of Pain During Stair-Climbing
NRS during stair-climbing | 3 months postoperatively
  Numeric Rating Scale of Pain During Stair-Climbing
NRS during stair-climbing | 1 year postoperatively
  Numeric Rating Scale of Pain During Stair-Climbing
NRS during stair-climbing | 2 years postoperatively
  Numeric Rating Scale of Pain During Stair-Climbing
NRS during performing sports | pre-operatively
  Numeric Rating Scale of Pain During Sports
NRS during performing sports | 3 months post-operatively
  Numeric Rating Scale of Pain During Sports
NRS during performing sports | 1 year post-operatively
  Numeric Rating Scale of Pain During Sports
NRS during performing sports | 2 years post-operatively
  Numeric Rating Scale of Pain During Sports
NRS during weight-bearing | pre-operatively
  Numeric Rating Scale of Pain During Weightbearing
NRS during weight-bearing | 3 months postoperatively
  Numeric Rating Scale of Pain During Weightbearing
NRS during weight-bearing | 1 year post-operativley
  Numeric Rating Scale of Pain During Weightbearing
FAAM | pre-operatively
  Foot and Ankle Ability Measure
FAAM | 3 months postoperatively
  Foot and Ankle Ability Measure
FAAM | 1 year postoperatively
  Foot and Ankle Ability Measure
FAAM | 2 years postoperatively
  Foot and Ankle Ability Measure
SF-12 | pre-operatively
  Short-Form 12
SF-12 | 3 months postoperatively
  Short-Form 12
SF-12 | 1 year postoperatively
SF-12 | 2 years postoperatively
  Short-Form 12
Ankle Activity Scale (AAS) | pre-operatively
Ankle Activity Scale (AAS) | 3 months postoperatively
Ankle Activity Scale (AAS) | 1 year post-operatively
Ankle Activity Scale (AAS) | 2 year post-operatively
Return to sports | post-operatively until 2 years of follow-up post-operatively
Return to work | post-operatively until 2 years of follow-up post-operatively
Radiological outcomes: CT-scan (depth, wide, length, joint space measurement) | pre-operatively
Radiological outcomes: CT-scan (depth, wide, length, joint space measurement) | 2 weeks postoperatively
Radiological outcomes: CT-scan (depth, wide, length, joint space measurement) | 1 year postoperatively
Radiological outcomes: CT-scan (depth, wide, length, joint space measurement) | 2 years postoperatively
Radiological outcomes: MRI scan (T2 relaxation times) | Pre-operatively
Radiological outcomes: MRI scan (T2 relaxation times) | 1 year post-operatively
Radiological outcomes: MRI scan (T2 relaxation times) | 2 years post-operatively
Cost-effectiviness | From per-operatively to post-operatively at 2 years (one period)
  all relevant clinical costs will be scored through a patient diary
Cell-subset analysis | per-operatively
  protein analyses will be performed by Sanquin
Demographic data | Pre-operatively
  all kinds of demographic data will be assessed (age, gender, etc.)
Complications | From per-operatively to post-operatively at 2 years (one period)
  all types of complications
Re-operations | From per-operatively to post-operatively at 2 years (one period)
  re-operations will be assessed

IPD SHARING:
Plan to Share IPD: Undecided